CLINICAL TRIAL: NCT00854906
Title: Comparison of Keratometric Tear Break Up Time (KTBUT) to Fluorescein Tear Break Up Time (FTBUT)
Brief Title: Keratometric Tear Breakup Time and Fluorescein Tear Breakup Time
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Richard Harper, MD, Department of Ophthalmology, University of Arkansas for Medical Sciences
Other Study IDs: 109338
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Dry Eye
Keywords: dry eye; keratometer; fluorescein
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Keratometric Tear Breakup Time: These are the study participants whose tear break up times were measured with a keratometer.
- Fluorescein Break Up Time: These are the study participants whose tear break up times were measured with with fluorescein dye.

SUMMARY:
The purpose of the research is to determine if putting fluorescein onto the eye (most common test done for dry eye syndrome) is an accurate way to measure dry eye symptoms. The investigators can avoid placing any foreign substance into the eye by using a manual keratometer. Therefore, the investigators want to compare the measurements of tear breakup time using fluorescein with using a novel method, a manual keratometer and then compare these measurements to a validated dry eye symptoms questionnaire. All qualifying patients who were scheduled in the Jones Eye Institute Clinics for a complete eye exam were offered information about the study and invited to participate. Participants were recruited from February 29, 2009 to April 14, 2009.Participants who did not meet the study protocol's inclusion and exclusion criteria were not included the study or study data analysis. All subjects eyes were measured for KTBUT and FTBUT.

DETAILED DESCRIPTION:
This is an observational study to measure the difference between Keratometric Tear Break Up Time (KTBUT) and Fluorescein Tear Break Up Time (FTBUT). All qualified study participants had their eyes measured for tear break up time measured with a keratometer and with fluorescein dye. In this study, we compare the use of the most common method, fluorescein dye, to measure tear break up time to a novel method, a keratometer, to measure tear break up time. Using the keratometer avoids instilling fluorescein dye into the tear film and not altering the tear film's physiologic environment.

ELIGIBILITY:
Inclusion Criteria:

* An adult, between ages 18-99
* An adult who is able to understand study instructions

Exclusion Criteria:

* An adult with corneal pathology that prevents accurate assessment of keratometric or fluorescein tear break up time.
* An adult with an allergy to fluorescein, a very common eye dye that detects defects in the cornea.
* The inability to answer questions on your own.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the Jones Eye Clinic, Department of Ophthalmology, University of Arkansas for Medical Sciences
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jones Eye Institute, University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All qualifying patients who were scheduled in the Jones Eye Institute Clinics for a complete eye exam were offered information about the study and invited to participate. Participants were recruited from February 29, 2009 to April 14, 2009.
Pre-assignment Details: Participants who did not meet the study protocol's inclusion and exclusion criteria were not included the study or study data analysis. All subjects eyes were measured for first for KTBUT and second for FTBUT. Each measurement occured three times in each eye and the results were recorded in seconds during their office visit and averaged.
Groups:
- All Study Participants: These are the total number of study participants whose tear break up times were measured with a keratometer (KTBUT) and fluorescein dye (FTBUT). Both KTBUT and FTBUT were measured in all study participants.
Period: Overall Study
Arm/Group | All Study Participants
Started | 26 (There were 26 participants whose eyes were measured in the KTBUT group.)
Completed | 25 (There were 26 participants in this group. One person was excluded be causes of no ocular history.)
Not Completed | 1
Not completed — One person had no ocular history | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: These are the total number of study participants whose tear break up times were measured with a keratometer (KTBUT) and fluorescein dye (FTBUT). All study participants participated in both the KTBUT Study Arm and the FTBUT Study Arm.
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Keratometric Tear Break Up Time (KTBUT) and Fluorescein Tear Break Up Time (FTBUT)
Description: This outcome measures the difference in tear break up time using a keratometer and fluorescein dye.
Time Frame: 1 day
Population: The number of participants for analysis was determined if each participant met all of the study protocol's inclusion and exclusion criteria. KTBUT and FTBUT were measured on all study participants.
Measure: Mean (Standard Deviation); unit: time in seconds
Units Other Than Participants: eyes
Arm/Group | KTBUT | FTBUT
Number analyzed (Participants) | 25 | 25
Number analyzed (eyes) | 50 | 50
time in seconds | 5.95 (2.8) | 5.39 (2.57)
Statistical Analysis 1: Comparison: KTBUT vs FTBUT; The paired T-test was used to compare mean KTBUT and mean FTBUT; Test type: Non-Inferiority or Equivalence — This was a pilot study. Therefore, no formal power analyses were performed; p = 0.074, t-test, 2 sided; Mean Difference (Final Values) = 0.666, 95% CI 2-sided [-0.069 to 1.401], Standard Deviation 3.6

2. Secondary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire
Description: The Ocular Surface Disease Index (OSDI) is a validated 12-item questionnaire used in dry eye studies. The OSDI Scale ranges from 0= Normal to 100= Severe. Subcategories include problems--all of the time, most of the time, half of the time,and none of the time.
Time Frame: 1 week
Population: By comparing the KTBUT and the FTBUT to the Ocular Surface Disease Index (OSDI) questionnaire score of each participant, we will be able to evaluate the difference in tear break up time using these items. The OSDI was given once before the participant's KTBUT and FTBUT was measured.
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
participants | 9.4 (9.1)
Statistical Analysis 1: Comparison: All Study Participants; A correlation was performed between ODSI questionnaire results and each participant's KTBUT; Test type: Non-Inferiority or Equivalence — The analysis will evaluate the association between OSDI with KTBUT; p = 0.093, Pearson's correlation; Pearson's Correlation, r = -0.34
Statistical Analysis 2: Comparison: All Study Participants; A correlation was performed between ODSI questionnaire results and each participant's FTBUT; Test type: Superiority or Other; p = 0.216, Pearson's Correlation; Pearson's Correlation, r = -0.26

ADVERSE EVENTS:
Description: The number of participants at risk were 0. Serious and/or other [non-serious] adverse events were not collected or assessed. The study only required subjects to participate one time. There were not any follow-up visits.
Arm/Group | KTBUT | FTBUT
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No